CLINICAL TRIAL: NCT04614337
Title: A Multicenter, 24-Month, Randomized, Open-Label, Active Control, Parallel Arm, Phase 2 Study of Daily Oral LUM-201 in Naïve-to-Treatment, Prepubertal Children With Idiopathic Growth Hormone Deficiency (GHD)
Brief Title: Phase 2 Study of LUM-201 in Children With Growth Hormone Deficiency (OraGrowtH210 Trial)
Acronym: OraGrowtH210
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lumos Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUM-201-01
Record Dates: First submitted 2020-10-26; First posted 2020-11-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Growth Hormone Deficiency
Keywords: GHD; Pediatric Growth Hormone Deficiency; LUM-201; Growth hormone secretagogue; Height; Catch-up growth; PEM; Oral; Predictive Enrichment Marker
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LUM-201 (0.8 mg/kg/day) (Experimental)
  Interventions: Drug: LUM-201
- LUM-201 (1.6 mg/kg/day) (Experimental)
  Interventions: Drug: LUM-201
- LUM-201 (3.2 mg/kg/day) (Experimental)
  Interventions: Drug: LUM-201
- rhGH (34 µg/kg/day) (Active Comparator)
  Interventions: Drug: rhGH Norditropin® pen (34 µg/kg)

INTERVENTIONS:
Drug: LUM-201 — Administered orally once daily
  Arms: LUM-201 (0.8 mg/kg/day); LUM-201 (1.6 mg/kg/day); LUM-201 (3.2 mg/kg/day)
Drug: rhGH Norditropin® pen (34 µg/kg) — Administered subcutaneously (s.c., under the skin) once daily.
  Arms: rhGH (34 µg/kg/day)

SUMMARY:
This is a multi-national trial. The goals of the trial are to study LUM-201 as a possible treatment for Pediatric Growth Hormone Deficiency (PGHD) and investigate a predictive enrichment marker (PEM) strategy to select subjects likely to respond to therapy with LUM-201.

DETAILED DESCRIPTION:
This trial will have one screening visit with tests to assess if subjects are eligible to start study therapy. Once subjects have completed screening, and if they are determined to be eligible, they will be randomized to receive one of three oral daily doses of LUM-201 or daily injections of recombinant human growth hormone (rhGH). All subjects will have an equal chance of being placed in any of the four groups.

The trial consists of up to 24 months of treatment. After screening, subjects will return to the clinic for 6 (subjects placed in rhGH group) or 10 visits (subjects placed in LUM-201 group). During several of these clinic visits, subjects will have a physical exam, blood, and urine collections. There will also be 3 phone calls with study staff that will take place between the clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Have an established diagnosis of idiopathic PGHD as determined by standard diagnostic criteria. Eligible subjects must be naïve-to-treatment and be prepubertal.
* Morning cortisol ≥ 7 µg/dL or stimulated cortisol ≥ 14 µg/dL.
* At Screening, be ≥ 3.0 years and ≤ 11.0 years for girls and ≤ 12.0 years for boys.
* Have HT-SDS ≤ -2.0 or HT-SDS ≥ 2 SD below mean parental HT-SDS.
* Have a baseline height velocity < 5.5 cm/year based on at least 6 months of growth.
* Have a bone age delayed by ≥ 6 months with respect to chronological age.
* Have prepubertal status as evidenced by Tanner Stage I breast development in girls and testicular volume < 4.0 mL in boys.
* In girls, have genetic testing results to rule out Turner syndrome. If SHOX genetic testing results are available, they need to be negative.
* Have normal thyroid function. Subjects diagnosed with hypothyroidism must have documented successful treatment for at least 30 days prior to Day 1.

Exclusion Criteria:

* Any medical or genetic condition which, in the opinion of the Investigator or Medical Monitor (MM), can be an independent cause of short stature and/or limit the response to exogenous growth factor treatment. (Examples: diabetes, idiopathic short stature).
* A medical or genetic condition that, in the opinion of the Investigator and/or MM, adds unwarranted risk to use of LUM-201 or rhGH.
* Use of any medication that, in the opinion of the Investigator and/or MM, can independently cause short stature or limit the response to exogenous growth factors (Example: glucocorticoids).
* Evidence or history of an intracranial mass (e.g., pituitary tumor, craniopharyngioma).
* Suspicion of absent pituitary function as evidenced by a maximal stimulated GH ≤ 3 ng/mL on two prior standard of care GH stimulation tests, or pituitary deficiencies beyond GH and thyroid function.
* Malnutrition as evidenced by medical history or a body weight < 3rdth percentile for current height.
* BMI > 95th percentile.
* Gestational age-adjusted birth weight < 5th percentile (small for gestational age).
* History of spinal, cranial, or total body irradiation.
* Treatment with medications known to act as moderate or strong inhibitors or strong inducers of CYP3A/4, or with medications known to act as strong inhibitors of P-glycoprotein (P-gp) or potent substrates of P-gp or Multidrug and toxin extrusion protein 1 (MATE1).

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects selected by PEM strategy who meet target growth | Day 1 to Month 6
  Annualized height velocity (AHV) measured as standing height with stadiometer
AHV after 6 months on LUM-201 compared to rhGH | Day 1 to Month 6
  Annualized height velocity to be measured

SECONDARY OUTCOMES:
Degree of concordance between the first and second assessment with the PEM strategy. | Screening to Day 1
  Peak serum concentration of GH in response to a single provocative dose of LUM-201
Incidence of adverse events in children with GHD | Day 1 to Month 24
  Number of events
Height standard deviation score (SDS) | Day 1 to Month 6 and Month 12
  Change in HT-SDS
Height velocity standard deviation score (HV-SDS) | Day 1 to Month 6, and Month 12
  Change in HV-SDS
Change in Weight | Day 1 to Month 6, and Month 12
  Change in Weight
Change in Weight SDS | Day 1 to Month 6 and Month 12
  Change in Weight-SDS
Change in BMI | Day 1 to Month 6 and Month 12
  Change in BMI
Change in BMI SDS | Day 1 to Month 6 and Month 12
  Change in BMI SDS
Bone Age | Day 1 to Month 6 and Month 18
  Change in bone age, measured by X-ray of left hand and wrist using Greulich & Pyle atlas
Pharmacokinetics of LUM-201 | Day 1 to Month 6 and 12
  Serum concentrations (Cmax/Steady State)
GH Concentration on maintenance treatment | Day 1 to Month 6 and 12
  Serum GH concentration
Insulin-like growth factor 1 SDS | Day 1 to Month 6 and 12
  Serum concentrations of insulin-like growth factor 1

CONTACTS AND LOCATIONS:
Locations (43):
- United States (27):
  - Center of Excellence in Diabetes and Endocrinology, Sacramento, California
  - Rady Children's Hospital, San Diego, California
  - Pediatric Endocrine Associates, Greenwood Village, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Novak Center For Childrens Health, Louisville, Kentucky
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - M Health, Fairview Pediatric Specialty Clinics- Discovery Clinic, Minneapolis, Minnesota
  - Children's Minnesota, Saint Paul, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - UBMD Pediatrics, Buffalo, New York
  - The Mount Sinai Hospital, Mount Sinai, New York
  - NYU Grossman School of Medicine, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Pediatric Diabetes and Endocrinology, Oklahoma City, Oklahoma
  - Penn State College of Medicine, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Tech University Health Sciences Center, Amarillo, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
- Australia (4):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Department of Pediatrics and Endocrinology- Monash Health, Clayton, Victoria
  - Royal Children's Hospital, Melbourne, Victoria
  - Queensland Children's Hospital, South Brisbane
- Schneider Children's Medical Center Institute for Endocrinology and Diabetes National Center, Petah Tikva, Tiqwa, Israel
- New Zealand (2):
  - Wellington Regional Hospital CCDHB, Newtown, Wellington Region
  - Liggins Institute, University of Auckland, Auckland
- Poland (8):
  - Klinika Pediatrii, Endokrynologii, Diabetologii z Pododdziałem Kardiologii, Uniwersytecki Dziecięcy Szpital Kliniczny im.Ludwika Zamenhofa w Białymstoku, Bialystok
  - Klinika Endokrynologii i Chorob Metabolicznych, Instytut Centrum Zdrowia Matki Polki, Lodz
  - Klinika Pediatrii, Diabetologii i Endokrynologii Gdansk, Pomorskie
  - klinika Pediatrii, Endokrynologii i Diabetologii Dziecięcej, Rzeszów
  - Sonomed - Centrum Medyczne, Szczecin
  - Klinika Endokrynologii i Diabetologii, Instytut "Pomnik Centrum Zdrowia Dziecka, Warsaw
  - SP Dziecięcy Szpital Kliniczny w Warszawie, Warsaw
  - Klinika Endokrynologii i Diabetologii Wieku Rozwojowego UM, Wroclaw
- State Institution 'V. P. Komissarenko Institute of Endocrinology and Metabolism of the National academy of medical science of Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided